CLINICAL TRIAL: NCT00970684
Title: A Phase II Study of Bevacizumab Plus Docetaxel and Gemcitabine in Subjects With Advanced, Previously Untreated, Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Bevacizumab, Docetaxel, and Gemcitabine Patients With Stage IIIB, Stage IV, or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nathan Pennell, MD, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Nathan Pennell, MD, PhD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4507; P30CA043703 (NIH); CASE4507 (Other: Case Comprehensive Cancer Center); CASE 4507-CC694 (Other: Cancer Center IRB); NCI-2010-00547 (Other: NCI/CTRP)
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2022-08-16 (Actual); Status verified 2022-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Bevacizumab; Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab, Docetaxel, and Gemcitabine (Experimental): Treatment repeats every 21 days for up to 6 courses.
  Interventions: Biological: bevacizumab; Drug: docetaxel; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Biological: bevacizumab — 15 mg/kg on day 1 of a 21-day cycle
Drug: docetaxel — 75 mg/m2 on day 1
Drug: gemcitabine hydrochloride — 900 mg/m2 on days 1, and 8,

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as docetaxel and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with docetaxel and gemcitabine hydrochloride may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with docetaxel and gemcitabine hydrochloride works in treating patients with stage IIIB, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the 1-year progression-free survival rate in patients with stage IIIB, stage IV, or recurrent non-squamous cell non-small cell lung cancer treated with bevacizumab, docetaxel, and gemcitabine hydrochloride.

Secondary

* Evaluate the median time to progression in patients treated with this regimen.
* Estimate the response rate in patients treated with this regimen.
* Determine the median overall survival of patients treated with this regimen.
* Determine the incidence of adverse events associated with this regimen in these patients.

OUTLINE: Patients receive bevacizumab IV over 30-90 minutes and docetaxel IV over 60 minutes on day 1 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with responsive or stable disease may then continue to receive bevacizumab alone for up to 12 months in the absence of disease progression.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-squamous cell non-small cell lung cancer

  * Stage IIIB (with pleural effusion), stage IV, or recurrent disease
* Bidimensionally measurable disease
* No known CNS disease, except for previously treated brain metastasis defined as no evidence of progression or hemorrhage after treatment AND no ongoing requirement for dexamethasone as documented by clinical examination, MRI, or CT scan

  * Treatment for brain metastases may have included whole brain radiotherapy, radiosurgery (gamma knife, LINAC, or equivalent), or a combination of therapy as deemed appropriate by the treating physician
  * Stable dose of anticonvulsants allowed
* No known metastatic disease to the gastrointestinal tract (e.g., stomach, small bowel, or large bowel)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 3 months
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Bilirubin ≤ 2.0 mg/dL
* AST or ALT ≤ 2.5 times upper limit of normal (ULN) (≤ 5.0 times ULN if hepatic metastases are present)
* Serum creatinine ≤ 1.8 mg/dL
* Urine protein:creatinine ratio < 1.0 OR proteinuria < 2+ by urine dipstick OR ≤ 1 g of protein by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Available for regular follow-ups
* No inadequately controlled hypertension, defined as systolic BP > 150 mm Hg and/or diastolic BP > 100 mm Hg despite antihypertensive medications
* No history of hypertensive crisis or hypertensive encephalopathy
* No NYHA class II-IV congestive heart failure
* No myocardial infarction or unstable angina within the past 6 months
* No stroke or transient ischemic attack within the past 6 months
* No significant vascular disease (e.g., aortic aneurysm, aortic dissection requiring surgical repair, or recent peripheral arterial thrombosis) within the past 6 months
* No symptomatic peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* No history of colonic diverticular disease (i.e., diverticulosis or diverticulitis)
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No serious, nonhealing wound, ulcer, or bone fracture
* No known hypersensitivity to any component of bevacizumab
* No hemoptysis (bright red blood of ≥ ½ teaspoon per episode) within the past 3 months
* No significant traumatic injury within the past 28 days

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or biological therapy
* No prior radiotherapy to an area of measurable disease unless there is documented progressive disease after completion of therapy
* More than 2 weeks since prior radiotherapy
* More than 4 weeks since prior and no concurrent participation in another experimental drug study, except for a Genentech-sponsored bevacizumab cancer study
* More than 28 days since prior major surgical procedure or open biopsy
* More than 3 months since prior abdominal surgery
* More than 3 months since prior neurosurgical resection or brain biopsy
* More than 7 days since prior core biopsy or other minor surgical procedure, except placement of a vascular access device
* No concurrent major surgical procedure

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Pennell, MD, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Afshin Dowlati, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Fairview Hospital, Moll Pavilion, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Hillcrest Hospital, a Cleveland Clinic Hospital, Mayfield Heights, Ohio

REFERENCES:
- [Derived] Patil PD, Shapiro M, Hashemi Sadraei N, Pennell NA. An Open-Label Phase II Trial of Bevacizumab plus Docetaxel and Gemcitabine in Advanced, Previously Untreated Nonsquamous Non-Small Cell Lung Cancer. Oncologist. 2019 Apr;24(4):457-e126. doi: 10.1634/theoncologist.2018-0857. Epub 2019 Jan 2. PMID 30602615

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from local medical clinics from 12/2009 to 4/2011
Period: Overall Study
Arm/Group | Bevacizumab, Docetaxel, and Gemcitabine
Started | 13
Completed | 3
Not Completed | 10
Not completed — Lack of Efficacy | 5
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab, Docetaxel, and Gemcitabine
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 63 [35 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival(PFS)
Description: PFS is defined as time to death or first occurrence of documented disease progression assessed by the investigator as per the RECIST guidelines (at lease a 20% increase in the diameter of a lesion, in addition to an absolute increase of 5mm). If no deaths occur prior to progression, this measure will be the same as the median time to progression.
Time Frame: 1 year
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab, Docetaxel, and Gemcitabine
Number analyzed (Participants) | 13
months | 5.6 [3.9 to 7.4]

2. Secondary Outcome: Median Time to Progression
Description: Time to progression (TTP) is defined as the time from start of treatment to first evidence of disease progression, defined per the RECIST 1.1 criteria as at least a 20% increase in the diameter of a lesion and an absolute increase of at least 5mm.
Time Frame: 1 year
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab, Docetaxel, and Gemcitabine
Number analyzed (Participants) | 13
months | 5.6 [3.9 to 7.4]

3. Secondary Outcome: Best Response
Description: The number of patients with a response will be assessed using the RECIST criteria of complete response (the disappearance of all target lesions); partial response (at least a 30% decrease in the diameter of lesions); progressive disease at least a 20% increase in the diameter of lesions); or stable disease(neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease)
Time Frame: 1 year
Population: One patient was unevaluable for response due to missing baseline tumor measurement.
Measure: Number; unit: participants
Arm/Group | Bevacizumab, Docetaxel, and Gemcitabine
Number analyzed (Participants) | 12
participants
  Stable Disease | 2
  Partial Response | 9
  Progressive Disease | 1

ADVERSE EVENTS:
Time Frame: Patients are followed for adverse events while on study for up to 2 years.
Arm/Group | Bevacizumab, Docetaxel, and Gemcitabine
Serious Adverse Events (participants affected / at risk) | 10/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab, Docetaxel, and Gemcitabine (N=13)
Anemia (Blood and lymphatic system disorders) | 1
Thromboembolic event (Vascular disorders) | 3
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Depressed Level of Consciousness (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab, Docetaxel, and Gemcitabine (N=13)
Allergic reaction/hypersensitivity (Immune system disorders) | 5 — including drug fever
Tinnitus (Ear and labyrinth disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Hemoglobinemia (Blood and lymphatic system disorders) | 10
Leukocytopenia (Blood and lymphatic system disorders) | 12
Lymphopenia (Blood and lymphatic system disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Superaventricular and nodal arrhythmia-Atrial fibrillation (Cardiac disorders) | 2
Supraventricular and nodal arrythmia-Sinus tachycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 2
Hypotension (Cardiac disorders) | 1
Fatigue (General disorders) | 10 — asthenia, lethargy, malaise
Fever (General disorders) | 2
Insomnia (General disorders) | 5
Rigors/chills (General disorders) | 1
Sweating (General disorders) | 3
Weight gain (General disorders) | 1
Weight loss (General disorders) | 6
Bruising (Skin and subcutaneous tissue disorders) | 1 — In absence of Grade 3 or 4 thrombocytopenia
Dry skin (Skin and subcutaneous tissue disorders) | 6
Flushing (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7
Nail changes (Skin and subcutaneous tissue disorders) | 4
Rash- acne/acneiform (Skin and subcutaneous tissue disorders) | 5
Ulceration (Skin and subcutaneous tissue disorders) | 2
Night Sweats, intermittent (Endocrine disorders) | 1
Anorexia (Gastrointestinal disorders) | 10
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Dehydration (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 8
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 3
Mucositis/stomatitis-oral (Gastrointestinal disorders) | 10
Mucositis/stomatitis-rectum (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Dysgeusia (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 6
Hemorrhage, GI (Gastrointestinal disorders) | 4
Hemorrhage-pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 7
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 3
Infection-Lung (Infections and infestations) | 4
Infection (Infections and infestations) | 6
Infection-Bladder (Infections and infestations) | 1
Infection-Conjuctiva (Infections and infestations) | 1
Infection-Mucosa (Infections and infestations) | 2
Infection-Upper aerodigestive NOS (Infections and infestations) | 1
Opportunistic infection (Infections and infestations) | 1 — associated with >= Grade 2 Lymphopenia
Edema-limb (Blood and lymphatic system disorders) | 3
Lymphocele (Blood and lymphatic system disorders) | 1
ALT, SGPT (Metabolism and nutrition disorders) | 4
AST, SGOT (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Alkaline phosphatase (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 12
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Glycosuria (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 5
Proteinuria (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Confusion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 4
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 2
Mood alterations (Nervous system disorders) | 6 — Anxiety/depression
Neuropathy (Nervous system disorders) | 8
Somnolence (Nervous system disorders) | 1
Dry eye syndrome (Eye disorders) | 1
Epiphora (Eye disorders) | 5
Pain- Abdomen NOS (Gastrointestinal disorders) | 1
Pain- Chest/thorax (Respiratory, thoracic and mediastinal disorders) | 3
Pain- dental/teeth/peridontal (General disorders) | 1
Pain- eye (Eye disorders) | 1
Pain- Head/headache (Nervous system disorders) | 6
Pain- Muscular/skeletal (Musculoskeletal and connective tissue disorders) | 9
Pain-other (General disorders) | 4
Pain- Throat/pharynx/larynx (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 — non-malignant
Pneumonititis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3
Sexual/reproductive function (Reproductive system and breast disorders) | 1
Thrombosis (Vascular disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes